CLINICAL TRIAL: NCT02621528
Title: Multi-center, Prospective, Post-market Study
Brief Title: Lifetech CeraFlex™ Post-Market Surveillance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CeraFlex™ PMSS
Record Dates: First submitted 2015-10-22; First posted 2015-12-03 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Patent Foramen Ovale; Atrial Septal Defect; Patent Ductus Arteriosus
Keywords: CeraFlex occluder
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Septal Defects, Atrial; Ductus Arteriosus, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CeraFlex occluder (Other): The Lifetech CeraFlex™ study is a triple-arm study.
  Interventions: Device: CeraFlex

INTERVENTIONS:
Device: CeraFlex — The Lifetech CeraFlex™ study is a triple-arm study.

SUMMARY:
The purpose of this multi-center, non-interventional, prospective, post-market clinical study is to collect real world data on patient outcomes and evaluate the procedural success and performance of the Lifetech CeraFlex™ occluders for patients with secundum type Atrial Septum Defect (ASD), Patent Foramen Ovale (PFO) or Patent Ductus Arteriosus (PDA).

DETAILED DESCRIPTION:
This study is designed as a post-market, prospective, multi-center, non-interventional clinical study to collect data regarding procedural success, clinical performance and cost-effectiveness of the Lifetech CeraFlex™ occluders in patients with secundum ASD, PFO and PDA.

Patients will be recruited in up to 12 investigational centers located in Europe and the Middle East.

To avoid bias in the study population the following measures will be taken:

* All sponsor or designee and external study personnel will be trained on the latest version of the Clinical Investigation Plan (CIP) and related study materials.
* Patients will be screened to confirm study eligibility with pre-defined inclusion/exclusion criteria prior to enrollment.
* This study will follow consecutive screening and enrollment.

The study will enroll 120 patients. The patient population will consist of up to approximately 40 consecutive enrolled patients with a confirmed secundum type ASD, up to approximately 40 enrolled patients with PFO and up to approximately 40 enrolled patients with PDA resulting in a significant shunt and in need of an intervention. These estimated upper limits per therapy group can however be exceeded depending on the enrollment trend, to account for a minimum of 10 patients to be enrolled per therapy group and a total study population of 120 enrolled patients.

ELIGIBILITY:
Inclusion criteria

To participate in this study, the patient must meet all of the following inclusion criteria:

1. Confirmed ASD, PFO or PDA and patient characteristics consistent with the corresponding IFU and sizing guidelines;
2. The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has signed the applicable Consent Form, approved by the appropriate Ethics Committee (EC)/IRB (where required);
3. The patient agrees to comply with requirements of the study including the 12 months followup.

Exclusion criteria

Patients will be excluded if any of the following conditions apply:

1. Any contra-indication mentioned in the corresponding IFU;
2. Currently participating in another investigational drug- or device study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Procedural success | immediate post procedure
  Absence of peri-procedural stroke/TIA, device embolization, cardiac or vascular perforation or death;Successful deployment of the occluder device(s).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Walsh, Professor, Principal Investigator — Our Lady's Children's Hospital, Crumlin
Locations (7):
- AP Hospital Europeen G Pompidou and Hospital Necker, Paris, France
- Germany (3):
  - Deutsches Herzzentrum Berlin, Berlin
  - Herzzentrum Leipzig GmbH, Leipzig
  - Deutsches Herzzentrum München, Munich
- Our Lady's Children's Hospital Crumlin, Dublin, Ireland
- Policlinico San Donato S.P.A., Milan, Italy
- Kinderspital Zürich, Zurich, Switzerland